CLINICAL TRIAL: NCT02533284
Title: Magnesium Sulfate for TAP Analgesia During Laparoscopic Cholecystectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, AlRefaey Kandeel, Dr, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 5
Record Dates: First submitted 2015-04-06; First posted 2015-08-26 (Estimated); Last update posted 2015-08-26 (Estimated); Status verified 2015-08

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Magnesium Sulfate; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Magnesium sulfate group (Experimental): US guided TAP with magnesium sulfate
  Interventions: Drug: Magnesium Sulfate; Drug: bupevecaine
- B group (Experimental): TAP bupevecaine
  Interventions: Drug: bupevecaine
- C group (Placebo Comparator): control TAP saline
  Interventions: Drug: saline

INTERVENTIONS:
Drug: Magnesium Sulfate — preemptive US guided TAP block will be done using Bupivacaine 0.25% plus 0.5 gm MgSo4 in M group).
  Other Names: Group 1
  Arms: Magnesium sulfate group
Drug: bupevecaine — US guided TAP using Bupevecaine 0.25 %
  Other Names: group 2
  Arms: B group; Magnesium sulfate group
Drug: saline — US guided TAP using placebo (saline)
  Other Names: group3
  Arms: C group

SUMMARY:
Study the effect of adding Magnesium sulfate to TAP block in analgesia after laparoscopic cholecystectomy.

DETAILED DESCRIPTION:
After approval of local ethical committee, consent will be obtained from 90 patients scheduled for laparoscopic cholecystectomy in GEC center, Mansoura University, Egypt. Patients will be of either ASA I and II, with Age ranging from 18-40 years, and BMI less than 35. Patients will be randomized into 3 groups (using closed envelope technique in blocks of 18); Controlled group (C group), Bupivacaine group (B group), Bupivacaine Magnesium group (M group).

Anesthesia induction will be the same in the three groups (Propofol 1-1.5mglkg, Fentanyl 1 mic/kg, Atracrium 0.5 mg/kg) then Sevoflorane inhalational anesthesia for maintainace in 0.4 oxygen/air mixtures.

In both M group and B group, preemptive US guided Subcostal TAP block (Toshiba Xario, Japan) was performed on both sides using 20 ml volume (0.25 Bupivacaine in B group or 0.25 Bupivacaine plus 0.5 gm MgSo4 in M group). Surgical sterilization will be started 5 minutes after the block and surgery started5 minutes later. Hemodynamic data (HR, MAP) will be collected immediately after induction, at start of surgery, and each 10 minutes later.

At the end of surgery, and after closure of surgical ports, anesthesia was terminated and extubation done when patients fulfilled the required criteria. Postoperative hemodynamic data (HR, MAP), VAS, and PONV will berecorded at 0, 1, 2, 6, 12, 24 hours after surgery, Ramsay sedation was recorded at 0, 1, 2, 6 hours postoperatively. Boluses of Morphine (0.02 mg/kg) will be given whenever VAS ≥4.

ELIGIBILITY:
Inclusion Criteria:

* ASA I, II for lap cholecystectomy

Exclusion Criteria:

* ASA III, IV

Ages: 16 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 90 (Estimated)
Dates: Start 2016-01; Primary Completion 2017-10 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
analgesia after laparoscopic cholecystectomy | 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura university, Al Mansurah, Dkahleya, Egypt